CLINICAL TRIAL: NCT05757050
Title: Evaluating the Effects of the Supplement ReFocus Tablets on Stress, Cognitive Function, Sleep and Wellbeing Following 14 Days Consumption in Healthy Volunteers Reporting Subjective Stress: A Randomised, Double-blind, Placebo Controlled, Crossover Trial
Brief Title: Mental Balance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A. Vogel AG (Industry)
Collaborators: University of Newcastle Upon-Tyne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5'000'750-1
Record Dates: First submitted 2023-02-15; First posted 2023-03-07 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Mental Health Wellness 1; Work Related Stress
MeSH Terms: conditions — Occupational Stress | interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Intervention Model Description: The proposed design is a randomised, double-blind, controlled, crossover intervention assessing the effects of an active intervention, containing Scutellaria baicalensis and Crataegus, versus placebo, on stress, cognition, sleep and wellbeing in healthy human volunteers. Outcome measures will be assessed acutely on day 1 and following 14 days of supplement consumption. Some interim outcome measures will also be assessed throughout the supplementation period to monitor sub-chronic changes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Re-Focus Tablets "Verum" (Experimental): The active intervention contains Scutellaria baicalensis (400 mg) and Crataegus (40 mg) and is in the form of a chewable tablet with a blood-orange flavour
  Interventions: Dietary Supplement: Re-Focus "Verum" Tablets; Dietary Supplement: Re-Focus "Placebo" Tablets
- Re-Focus Tablets "Placebo" (Placebo Comparator): The placebo will be a matched control
  Interventions: Dietary Supplement: Re-Focus "Verum" Tablets; Dietary Supplement: Re-Focus "Placebo" Tablets

INTERVENTIONS:
Dietary Supplement: Re-Focus "Verum" Tablets — The active intervention contains Scutellaria baicalensis (400 mg) and Crataegus (40 mg) and is in the form of a chewable tablet with a blood-orange flavour
  Other Names: Verum
Dietary Supplement: Re-Focus "Placebo" Tablets — The placebo will be a matched control.
  Other Names: Placebo

SUMMARY:
The proposed design is a randomised, double-blind, controlled, crossover intervention assessing the effects of an active intervention, containing Scutellaria baicalensis and Crataegus, versus placebo, on stress, cognition, sleep and wellbeing in healthy human volunteers. Outcome measures will be assessed acutely on day 1 and following 14 days of supplement consumption. Some interim outcome measures will also be assessed throughout the supplementation period to monitor sub-chronic changes

DETAILED DESCRIPTION:
Participants will attend the laboratory on 5 occasions. The first visit will take place on day -2 (this is a minimum period and can take place a maximum of 14 days prior to the baseline lab visit. A training refresher will take place if 14 days is exceeded) and represents an in-person screening and training visit. (This takes place following an earlier telephone pre-screen where participants will confirm that they meet the study inclusion criteria, and not any of the exclusion criteria (performed separately, this refines the lab-based screening/training visit).) Here participants will provide written, informed consent, complete demographic and anthropometric measurements (BMI & WHR) and be trained on the COMPASS cognitive tasks and study questionnaires.

If progressed through training/screening, participants will then return to the lab, on day 1, to complete their baseline lab visit for arm 1. This will take place at approximately 10:00 am, with participants having consumed their normal breakfast no later than 8:30 am that morning. Participants will first complete the PROM questionnaires and a baseline GSR reading (including a day-baseline saliva sample) will also be taken during this time. For the next 50 minutes, participants will complete the pre-dose COMPASS cognitive task battery and, after a short break, participants will complete the pre-dose OMS. At approximately 11:50 am, participants will consume their full daily treatment dose (2 tablets) along with a standardised lunch of a white bread cheese sandwich, packet of ready salted crisps, and a custard pot. After an hour-long 'absorption' period, participants will complete the post-dose COMPASS cognitive tasks and OMS and the testing day will be completed at approximately 2:30 pm.

Before leaving the lab, participants will be provided with their 14 (+/- the additional doses required for compliance and in case of delayed return for the chronic visit) days-worth of treatment, alongside a treatment diary to note down the time of treatment consumption each day. (The number of returned tablets on day 15, alongside reference to this treatment diary, will serve as the study compliance measures.) Participants will be advised to adhere to the following dosing regimen for each day going forward; 1 tablet in the morning, 1 in the evening, to be consumed 1 hour away from meals. On day 7 (+/- 2 days), participants will complete the PROM questionnaires, via survey, at home.

Participants will return to the lab on day 15 (+/- 2 days), following 14 full days of treatment, for the chronic lab visit for arm 1, and repeat the same procedure as day 1. A minimum 14-day washout period (with a maximum of 28 days) will then commence.

On day 30, participants will return to the lab for the baseline visit for arm 2 and repeat the same procedure as the acute arm 1 for visit. During the interim period, treatment will be consumed in the same way and, half-way through the dosing period (day 36 (+/- 2 days)) participants will complete the PROM questionnaires, via survey, at home.

On day 44 (+/- 2 days) participants will return to the lab for the chronic lab visit for arm 2, their final visit, which will be identical to the arm 1 chronic lab visit, with the exception that participants will be debriefed at the end of their visit and participant payment arranged. Here, participants will also be asked which treatment order they believed themselves to be on.

Please see figure 3 for the overall trial diagram and figure 4 for the procedure within the acute and chronic testing sessions.

ELIGIBILITY:
Inclusion Criteria:

* 18-75

Exclusion Criteria:

* • If participant scores less 12, or less, on the Perceived Stress Scale

  * Have any pre-existing medical condition/illness which will impact taking part in the study

    * NOTE: the explicit exceptions to this are controlled hyper/hypothyroidism, hay fever, high cholesterol and reflux-related conditions
  * Are currently taking prescription medications

    *NOTE: the explicit exceptions to this are contraceptive treatments for female participants, thyroid medications, topical skin treatments and those medications used in the treatment of high cholesterol and reflux-related conditions; and those taken 'as needed' in the treatment of asthma and hay fever
  * Have high blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg). NOTE: that we must measure this in the lab using our blood pressure monitors and can only use our measurements to assess eligibility rather than home or GP readings
  * Have a Body Mass Index (BMI) outside of the range 18.5-35 kg/m2
  * Are pregnant, seeking to become pregnant or lactating
  * Have learning and/or behavioural difficulties such as dyslexia or ADHD
  * Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour-blindness)
  * Smoke tobacco or vape nicotine or use nicotine replacement products (if you have recently quit smoking or using replacements you must have stopped using them altogether for a period of 3 months before participating in this study)
  * Have excessive caffeine intake (>500 mg per day). Note: This will be calculated at screening but feel free to query this with the researcher prior to attendance
  * Have relevant food allergies/ intolerances/ sensitivities (Please discuss with researcher prior to attendance if you are unsure of relevance)
  * Have taken antibiotics within the past 4 weeks
  * Have taken dietary supplements e.g. vitamins, omega 3 fish oils etc. in the last 4 weeks (Note: participation is possible following a 4-week supplement washout prior to participating and for the duration of the study on the proviso that the supplements are taken are out of choice and are not medically prescribed or advised). Existing and consistent use of vitamin D supplements and protein shakes are permitted
  * Have any health condition that would prevent fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)
  * Are unable to complete all of the study assessments
  * Are currently participating in other clinical or nutrition intervention studies, or have in the past 4 weeks
  * Have been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months
  * Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months, including a medical diagnosis of anxiety or depression.
  * Suffers from frequent migraines that require medication (more than or equal to 1 per month)
  * Have oral disease
  * Have any known active infections
  * Does not have a bank account (required for payment)
  * Are non-compliant with regards treatment consumption

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive function - Cognitive domain factor score | Prior to (baseline) and chronic (2 weeks) of intervention
  Speed of attention, accuracy of attention, speed of memory, accuracy of working memory, and accuracy of episodic memory measured by Computerised Mental Performance Assessment System (COMPASS, Northumbria University)
Change in Cognitive function - Cognitive domain factor score | Prior to (baseline) and following acute (60 minutes post-dose) of intervention
  Speed of attention, accuracy of attention, speed of memory, accuracy of working memory, and accuracy of episodic memory measured by Computerised Mental Performance Assessment System (COMPASS, Northumbria University)

SECONDARY OUTCOMES:
Profile of Mood States (POMS) | Prior to (baseline) and following 1 and 2 weeks of intervention
  35-item measure, summed to create measures of vigour, tension, fatigue, depression, confusion, anger, friendliness and total mood disturbance
Perceived Stress Scale (PSS) | Prior to (baseline) and following 1 and 2 weeks of intervention
  10-item measure, summed to create a single value with higher scores indicating higher levels of stress
State-Trait Anxiety Inventory (STAI) - Trait subscale | Prior to (baseline) and following 1 and 2 weeks of intervention
  20 item measure, summed to create a measure of trait anxiety
World Health Organisation Quality of Life Questionnaire (WHOQOL-BREF) | Prior to (baseline) and following 1 and 2 weeks of intervention
  World Health Organisation Quality of Life Questionnaire (WHOQOL-BREF)
Subjective sleep continuity | Prior to (baseline) and following 1 and 2 weeks of intervention
  Perceived sleep continuity as assessed by subjective sleep diary (measuring: Sleep latency, time in bed, number of awakenings, wake after sleep onset, total sleep time, sleep efficiency, nocturnal physical tension, nocturnal psychological tension, sleep enjoyment and feelings of restedness)
Subjective sleep via Patient-Reported Outcome Measurement, Information System Sleep Disturbance scale (PROMIS-SD) | Prior to (baseline) and following 1 and 2 weeks of intervention
  8-item measure, summed to create a single value with higher scores indicating higher levels of sleep disturbance
Depression, Anxiety and Stress scale (DASS-21) | Prior to (baseline) and following 1 and 2 weeks of intervention
  21 item measure, summed to create 3 component scores; depression, anxiety and stress.
Visual Analogue Mood Scales (VAMS) | Prior to (baseline) and following 1 and 2 weeks of intervention
  18 visual analogue scales scored along a 100 mm line, combined to give an average score on 3 factors: Alertness, Tranquillity and Stress
Visual Analogue Scales (VAS) | Prior to (baseline) and following 1 and 2 weeks of intervention
  Visual analogue scales scored along a 100 mm line, including 'relaxed', 'stress', 'anxious', 'calm'
Cognitive function - Individual cognitive task score | Prior to (baseline) and following acute (60 minutes post-dose) and chronic (2 weeks) intervention
  Individual tasks include the following: Immediate word recall, numeric working memory, choice reaction time, Corsi blocks, Peg and ball, delayed word recall, delayed word recognition, delayed name to face recall, delayed picture recognition measured by COMPASS, Northumbria University
Cognitive function - Cognitively demanding tasks | Prior to (baseline) and following acute (60 minutes post-dose) and chronic (2 weeks) intervention
  Cognitive function and mental fatigue during extended performance of cognitively demanding tasks (Cognitive Demand Battery, comprising serial 3s subtractions, serial 7s subtractions, rapid visual information processing task, and mental fatigue scale, repeated 3 times). Measured COMPASS, Northumbria University
Subjective stress reactivity - State-Trait Anxiety Inventory (STAI), State subscale | Prior to (baseline) and following acute (120 minutes post-dose) and chronic (2 weeks) intervention
  20 item measure, summed to create a measure of subjective state anxiety. Measured as response to psychological stressor
Physiological stress reactivity - cortisol and a-amylase | Prior to (baseline) and following acute (120 minutes post-dose) and chronic (2 weeks) intervention
  Measuring salivary cortisol and a-amylase to determine response to psychological stressor
Physiological stress reactivity - Galvanised skin response (GSR) | Prior to (baseline) and following acute (120 minutes post-dose) and chronic (2 weeks) intervention
  Measuring galvanised skin response to psychological stressor
Physiological stress reactivity - Heart rate (HR) | Prior to (baseline) and following acute (120 minutes post-dose) and chronic (2 weeks) intervention
  Measuring heart rate in response to psychological stressor
Cognitive function during psychological stressor | Prior to (baseline) and following acute (120 minutes post-dose) and chronic (2 weeks) intervention
  Individual tasks include the following: serial 3s subtractions, serial 7s subtractions, serial 17s subtractions and a tracking task during psychological stressor
Visual Analogue Mood Scales (VAMS) | Prior to (baseline) and following one dose (acute) at 60 minutes post-dose
  18 visual analogue scales scored along a 100 mm line, combined to give an average score on 3 factors: Alertness, Tranquillity and Stress
Visual Analogue Scales (VAS) | Prior to (baseline) and following one dose (acute) at 60 minutes post-dose
  Visual analogue scales scored along a 100 mm line, including 'relaxed' 'stress' 'anxious' 'calm'

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne & Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pseudonymized and compiled data sheets only

REFERENCES:
- [Derived] Dodd F, Weishaupt R, Katumba PKM, Elcoate R, Wightman E. Effects of a Scutellaria baicalensis/Crataegus laevigata, magnesium and chromium supplement on stressed individuals: A randomised, double-blind, placebo-controlled, crossover trial. J Psychopharmacol. 2025 Dec;39(12):1420-1436. doi: 10.1177/02698811251381261. Epub 2025 Nov 5. PMID 41194549